CLINICAL TRIAL: NCT00270361
Title: Management of Patients With CHF After Hospitalization-Follow up Serial Infusions of NATRECOR (Nesiritide) - FUSION I, A Pilot Study
Brief Title: FUSION I Assesses Safety and Tolerability of Two Doses of NATRECOR (Nesiritide) Administered to Patients With Worsening Congestive (Decompensated) Heart Failure Who Are Concurrently Receiving Their Usual Cardiac Medications and Are at High Risk for Hospitalization.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003316; NATRECORHFA2001; NCT00040612 (obsolete NCT alias)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; Renal Dysfunction; Cardiomyopathy; Heart Decompensation; Dyspnea Paroxsymal; Outpatient Therapy.
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardiomyopathies | interventions — Natriuretic Peptide, Brain

ARMS (3):
- 001 (Experimental): nesiritide
  Interventions: Drug: nesiritide
- 002 (Experimental): nesiritide
  Interventions: Drug: nesiritide
- 003 (Active Comparator): usual long term cardiac medications
  Interventions: Drug: usual long term cardiac medications

INTERVENTIONS:
Drug: nesiritide
  Arms: 001
Drug: usual long term cardiac medications
  Arms: 003
Drug: nesiritide
  Arms: 002

SUMMARY:
The purpose of this study is to assess the safety and tolerability of two doses of nesiritide (a recombinant form of the natural human peptide normally secreted by the heart in response to heart failure) when administered serially as a treatment to outpatients with worsening congestive heart failure (decompensated CHF) who are receiving their usual cardiac medications and are at high risk for hospitalization.

DETAILED DESCRIPTION:
Efforts to contain rising costs for hospital acute care have resulted in shorter hospital stays for patients with acutely decompensated heart failure. These shorter stays may not allow for adequate diuresis, titration of oral medications, or for patients to receive the full benefit of intravenously (IV) administered medications. In addition to shorter stays when hospitalized, physicians are exploring ways to treat patients in the outpatient setting to avoid hospitalization. Although there is increasing interest among clinicians in the use of outpatient IV therapy for the treatment of advanced heart failure, there is no consensus among clinicians regarding patient selection, dosing, or treatment duration. The use of IV inotropic agents (drugs that influence and or affect muscle contractility) such as milrinone or dobutamine in this setting is controversial and may lead to increased mortality. Indeed, the ACC/AHA (American College of Cardiology and American Hospital Association) guidelines warn that long-term intermittent use of IV inotropes for treatment of left ventricular dysfunction is of "unproved value and not recommended." Yet, despite these guidelines, clinicians use inotropes in the outpatient setting because there is no currently approved alternative therapy. Thus, there is an unmet need for effective outpatient treatment of advanced chronic heart failure to improve quality of life and/or reduce the number of hospital admissions for heart failure.

The data from previous studies suggest that doses of NATRECOR® hBNP may be a potent agent for the treatment of acute congestive heart failure (CHF) with a unique combination of desirable effects on the flow of blood throughout the body; the hormones secreted by the nervous system and support of copious salt outputs by the renal system not provided by currently available therapies. This study is a multicenter, open-label pilot study in which subjects who have received treatment for acutely decompensated CHF during a hospitalization at least twice within the previous 12 months are randomized (1:1:1) to one of three treatment groups. One treatment group will receive their usual long term cardiac medications, either with or without serial infusions of inotropes (various drugs that affect the strength of contractions of the heart muscle) and without nesiritide therapy. The 0.005 mcg/kg/min nesiritide treatment group receives a 0.5 mcg/kg bolus of nesiritide followed by a 0.0025 mcg/kg/min infusion, in addition to their usual long term cardiac medications, excluding IV inotropes; The 0.010 mcg/kg/min nesiritide treatment group receives a 1 mcg/kg bolus of nesiritide followed by a 0.005 mcg/kg infusion, in addition to their usual long term cardiac medications, excluding IV inotropes. Because patients treated in an outpatient setting may be less decompensated than patients with acutely decompensated heart failure, this study was designed to evaluate the 0.010 mcg/kg/min dose of nesiritide (the currently approved dose for acutely decompensated patients) as well as a lower dose (0.005 mcg/kg/min).

The hypothesis is that as an adjunct therapy to oral medications, serial IV infusions of nesiritide may produce more rapid and sustained compensation of heart failure in patients with frequent episodes of decompensated heart failure. The 0.005 mcg/kg/min group receives a 0.5 mcg/kg bolus followed by a 0.0025 mcg/kg/min infusion; the 0.010 mcg/kg/min group receives a 1 mcg/kg bolus followed by a 0.005 mcg/kg infusion. Intravenous bolus over 60 seconds and a fixed rate infusion of 4 - 6 hours, at least once per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having had at least two hospital admissions (or equivalent treatment) for acutely decompensated CHF within the last 12 months, with at least one of these admissions in the past 30 days, and having received treatment with intravenous vasoactive agents (such as intravenous inotropes, NATRECOR®, or nitroglycerin)
* able to be enrolled and initiate treatment with study drug within 5 to 30 days of last hospital discharge (or equivalent treatment) of acutely decompensated CHF
* have a baseline NYHA (New York Heart Association) Functional Classification III or IV for at least 2 months prior to randomization
* currently receiving optimal treatment with long term oral medications (e.g., diuretics, ACE inhibitors, and beta blockers, unless beta blockers or ACE inhibitors are documented to be contraindicated or not tolerated)
* willing to receive infusions of NATRECOR®, or possibly other medications, at least as frequently as once per week for 12 weeks.

Exclusion Criteria:

* Subjects having systolic blood pressure consistently less than 90 mm Hg
* having had organ transplantation (heart, liver, lung and kidney) in the past or anticipating organ transplantation during the study
* not able or willing to discontinue intermittent or continuous infusions of inotropes if randomized to a NATRECOR® treatment group
* having had a bi-ventricular pacemaker placed within the past 60 days or an automatic implantable cardiac defibrillator placed within the past 30 days
* requiring chronic dialysis or have an expectation that dialysis will be required during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2001-12; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment of nesiritide as an adjunct to standard medical therapy

SECONDARY OUTCOMES:
In NYHA Class IV patients with renal disease; number of hospitalizations, deaths, adverse cardiovascular events, and, adverse renal events

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Yancy CW, Saltzberg MT, Berkowitz RL, Bertolet B, Vijayaraghavan K, Burnham K, Oren RM, Walker K, Horton DP, Silver MA. Safety and feasibility of using serial infusions of nesiritide for heart failure in an outpatient setting (from the FUSION I trial). Am J Cardiol. 2004 Sep 1;94(5):595-601. doi: 10.1016/j.amjcard.2004.05.022. PMID 15342289